CLINICAL TRIAL: NCT01479179
Title: Phase I/II Study of Trastuzumab in Combination With AMG 479, A Fully Human Monoclonal Antibody Against Insulin-Like Growth Factor Type 1 Receptor (IGF-1R), in Patients With HER-2 Overexpressing Metastatic Breast Cancer Progressing on Trastuzumab-Based or Lapatinib-based Therapy
Brief Title: Trastuzumab in Combination With AMG 479 in HER-2 Overexpressing MBC Progressing on Trastuzumab
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Drug sponsor decision to discontinue study.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0542
Record Dates: First submitted 2011-11-21; First posted 2011-11-24 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Metastatic Breast Cancer; HER-2-overexpressing breast cancer; Human epidermal growth factor receptor; AMG 479; Trastuzumab; Herceptin
MeSH Terms: conditions — Breast Neoplasms | interventions — ganitumab; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AMG 479 + Trastuzumab (Experimental): AMG 479 18 mg/kg or 12 mg/kg intravenously (IV) 30 minutes after trastuzumab. Trastuzumab loading dose (Week 1) 8 mg/kg IV over 90 minutes; maintenance dose 6 mg/kg IV over 30 minutes every 3 weeks.
  Interventions: Drug: AMG 479; Drug: Trastuzumab

INTERVENTIONS:
Drug: AMG 479 — Phase I Starting Dose: 18 mg/kg by vein on Day 1 of a 21 day cycle.
  Phase II Starting Dose: Maximum tolerated dose from Phase I.
Drug: Trastuzumab — Phase I and II Starting Dose: 8 mg/kg by vein on Day 1 of a 21 day cycle.
  Phase I and II Maintenance Dose: 6 mg/kg by vein on Day 1 of a 21 day cycle.
  Other Names: Herceptin

SUMMARY:
The goal of Phase 1 of this clinical research study is to test the safety and tolerability of AMG 479 when given with trastuzumab.

The goal of Phase 2 of this clinical research study is to learn if the combination of AMG 479 and trastuzumab can help to control breast cancer.

AMG 479 is designed to block tumor cells from growing and spreading.

Trastuzumab is designed to prevent or slow down the growth of cancer cells by blocking proteins inside the cancer cell.

DETAILED DESCRIPTION:
Phase 1 and Phase 2 of the Study:

If you are found to be eligible to take part in this study, you will be assigned to a study group based on when you join this study. Groups of 3 participants will be enrolled in the Phase 1 portion of the study. There are 2 dose levels that will be tested in Phase 1.

If you are enrolled in the Phase 1 portion, the dose of AMG 479 you receive will depend on when you joined this study. The first group of participants will receive the higher dose level of AMG 479. If there are intolerable side effects, the next group will receive the lower dose.

If you are enrolled in the Phase 2 portion, you will receive AMG 479 at the highest dose that was tolerated in the Phase 1 portion.

All participants will receive the same dose level of trastuzumab.

Study Drug Administration:

You will receive AMG 479 by vein over 60-120 minutes on Day 1 of each 21-day cycle.

You will receive trastuzumab by vein over 30-90 minutes on Day 1 of each cycle.

If you are already receiving trastuzumab at the time you join the study, you will continue to receive the standard dose of trastuzumab. If the last dose of trastuzumab was given more than 1-3 weeks before you joined the study (depending on the dose previously received), then you will receive a higher "loading" dose of trastuzumab followed by the standard dose.

Study Visits:

At every visit, you will be asked about any side effects you may have had.

Your vital signs will be checked before, during, and after each infusion of AMG 479.

On Day 1 of Cycle 1, blood (about 5 tablespoons) will be drawn for routine tests.

If you are in Phase 1, blood (about 1 tablespoon each time) will be drawn for pharmacokinetic (PK) testing 2 times (before and after the study drug dose) on Day 1 of Cycles 1 and 2. PK testing measures the amount of study drug in the body at different time points.

On Day 8 of Cycle 1, blood (about 1 tablespoon) will be drawn for routine tests.

On Day 15 of Cycle 1:

* You will have a physical exam, including measurement of your weight and vital signs.
* Blood (about 1 tablespoon) will be drawn for routine tests.
* Your performance status and any updates to your medical history will be recorded.

On Day 1 of Cycles 2, 4, and 6, you will have CT or MRI scans to check the status of the disease.

On Day 1 of Cycles 2 and beyond:

* Blood (about 1-2 teaspoons) will be drawn for blood sugar tests. You will need to fast for 8 hours before these tests.
* You will have a physical exam, including measurement of your weight and vital signs.
* Your performance status and any updates to your medical history will be recorded.
* Blood (about 1 tablespoon) will be drawn for routine tests.

You will have a PET-CT scan at Week 3 if you had a PET-CT scan at screening.

On Day 8 of Cycles 1-3, blood (about 1½ teaspoons) will be drawn to check your blood clotting function.

Every 3 months, you will have either an ECHO or MUGA scan to check your heart function.

In certain cases with your doctor's permission, the study visits may occur 1 day earlier or later than described above. If you are having side effects, extra clinic visits may be needed.

Length of Treatment:

You may continue taking the study drugs for as long as the doctor thinks it is in your best interest. You will no longer be able to take the study drugs if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation on the study will be over once you have completed the end-of-treatment visit.

End of Treatment Visit:

Within 30 days after the last study drug dose:

* You will have a physical exam, including measurement of your weight and vital signs.
* You will be asked if you have had any side effects and about any drugs you may be taking.
* Any updates to your medical history will be recorded.
* Blood (about 3 tablespoons) will be drawn for routine tests.
* You will have a hearing test
* If you have not had one in the last 30 days or after your last treatment, you will have an ECHO or MUGA scan to check your heart function.
* If the doctor thinks it is needed, you will have CT or MRI scans to check the status of the disease.
* If you are in Phase 1, blood (about 1 tablespoon) will be drawn for PK testing.

This is an investigational study. Trastuzumab is FDA approved and commercially available for the treatment of breast cancer. AMG-479 is not FDA approved or commercially available. AMG-479 is currently being used for research purposes only.

Up to 35 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. History of biopsy-proven HER-2-overexpressing breast cancer and radiographic evidence of metastatic disease. The HER-2 status can be determined either by immunohistochemistry (score, 3+) or by fluorescence in situ hybridization.
2. Patients must have received anthracycline-, taxane- and capecitabine-based chemotherapy for breast cancer. In addition, patients must have developed progressive disease to trastuzumab- or lapatinib-based therapy within the last 3 months. Patients who develop metastatic breast cancer within 3 months after receiving trastuzumab or lapatinib in the adjuvant and/or neoadjuvant setting are eligible. Three prior lines of HER2-directed therapy (containing either trastuzumab or lapatinib) for metastatic breast cancer are allowed.
3. Woman >/=18 years old.
4. Performance status 0-2 (by Eastern Cooperative Oncology Group {ECOG} scale).
5. Laboratory parameters: Absolute neutrophil count (ANC) 1.0 x 10^9/L or higher; Platelet count 100,000 x 10^9/L or higher; Hemoglobin 9.0 g/dL or higher; Partial thromboplastin (PTT) </= 1.3 x upper limit of normal (ULN) and international normalized ratio (INR) </= 1.5, unless subject is on anticoagulation therapy. Subjects on therapeutic anticoagulation are eligible if there is no bleeding and they are on a stable dose of anticoagulation therapy (eg, on coumadin with an INR of 2 to 3) for at least 7 days before registration(prior to the start of therapy). Continued in inclusion #6.
6. Continuation from # 5: Serum creatinine </= 1.5 x the ULN or calculated creatinine clearance (by Cockcroft-Gault formula) >/=40 mL/min; Aspartate aminotransferase (AST) </= 2.5 x ULN; Alanine aminotransferase (ALT) </= 2.5 x ULN; Alkaline phosphatase </= 2.5 x ULN (</= 5 x ULN with bone/liver metastases ); Bilirubin </= 1.5 x ULN.
7. Glycosylated hemoglobin (HgbA1c)</= 8%
8. Fasting blood glucose </= 160 mg/dL (Fasting will require subjects to refrain from all food and beverage [except water] for at least 8 hours). Documentation will confirm patient compliance with nothing by mouth (NPO) status prior to lab exam.
9. Patients must not be pregnant. A pregnancy test will be obtained if the patient is a woman of child-bearing potential, defined as a sexually mature woman who has not undergone a hysterectomy or who has not been naturally postmenopausal for at least 24 consecutive months (i.e., who has had menses at any time in the preceding 24 consecutive months).
10. Patients must have signed an informed consent document stating that they understand the investigational nature of the proposed treatment.
11. Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >/= 20 mm with conventional techniques, including palpation, plain x-ray, or magnetic resonance imaging (MRI), or or >/= 10 mm with spiral computed tomography (CT) scan. Bone metastases and pleural effusions are not considered measurable disease.
12. Patients may not be receiving any other investigational agents within 30 days of registration.
13. Left ventricular ejection fraction determined by echocardiogram or multiple-gated acquisition scan (MUGA) (cardiac scan) must be 50% or higher.

Exclusion Criteria:

1. Central nervous system (CNS) metastases , unless previously treated by either radiation therapy and/or surgical resection, clinically stable and off corticosteroids. Subjects with a history of CNS metastases that are both treated and stably controlled are eligible if all of the following apply: therapy has been administered (surgery and/or radiation therapy); there is no additional treatment planned for brain metastases; the subject is clinically stable; the subject is off corticosteroids or on a stable dose of corticosteroids for at least 14 days prior to enrollment
2. Prior malignancy (other than in situ cervical cancer, or basal cell or squamous cell carcinoma of the skin), unless treated with curative intent and without evidence of disease for 3 years or longer.
3. Administration of other prior anticancer therapies within 4 weeks of enrollment, except Trastuzumab and Lapatinib.
4. Toxicities related to prior anticancer treatment (except alopecia) that have not resolved to </= grade 1 according to common terminology criteria for adverse events (CTCAE V4.0) before registration or prior to start of therapy.
5. Prior treatment with investigational treatment targeted to IGF axis including, but not limited to, CP-751,871, IM-A12, RO4858696.
6. Previous exposure to AMG 479.
7. Currently receiving systemic antibiotic therapy for the treatment of an active infection.
8. History of bleeding diathesis.
9. Known positive test for human immunodeficiency virus, or chronic hepatitis B or C infection.
10. Any co-morbid medical condition that may put the subject at significant risk for toxicity.
11. Major surgical procedure within 28 days of registration (prior to the start of therapy).
12. Minor surgical procedures within 7 days of registration although placement of central access device, fine needle aspiration, thoracentesis or paracentesis > 1 day before registration is acceptable.
13. Known inability to tolerate intravenous (IV) drug administration.
14. Has not yet completed at least 30 days before registration since ending other investigational device or drug study(s)
15. Subject has known sensitivity to any of the products to be administered during dosing.
16. Subject will not be available for follow-up assessments.
17. Subject has any kind of disorder that compromises the ability of the subject to give written informed consent and/or to comply with study procedures.
18. Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
19. History of venous thromboembolism.
20. Patient with reproductive potential who will not agree to use one highly effective method of contraceptive such as implants, injectables, intrauterine devices (IUDs) such as copper T or Levonorgestrel-releasing intrauterine system (LNG-IUS), sexual abstinence, vasectomised partner, or condom or occlusive cap (diaphragm or cervical/vault cap) supplemented with the use of a spermicide during treatment.
21. Poorly controlled diabetes mellitus
22. Patient with hearing impairment of > grade 3.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-11; Primary Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | After first 21 day cycle
  Maximum tolerated dose (MTD) is highest dose for which one or fewer dose limiting toxicities (DLTs) are experienced in 6 participants. DLT is defined as a grade 3, or higher hematological or non-hematological toxicity related to study (AMG-479) drug or combination of AMG 479 and trastuzumab therapy during first cycle (21 days).

SECONDARY OUTCOMES:
Clinical Benefit Rate (CBR) | Baseline to 24 weeks
  Efficacy measured by clinical benefit rate {CR (Complete response) + PR (Partial response) + SD (stable disease) >/= 24 weeks}. Response assessment by CT or MRI. CR: Disappearance of all target lesions; PR: >30% decrease in sum of longest diameter (LD) of target lesions, reference baseline sum LD; PD: =/>20% increase in sum of LD of target lesions, reference smallest sum LD recorded since treatment started or appearance of 1 or > new lesions. SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, reference smallest sum LD since treatment started.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco J. Esteva, MD,PHD, Principal Investigator — UT MD Anderson Cancer Center

REFERENCES:
- See also: UT MD Anderson Cancer Center — https://www.mdanderson.org